CLINICAL TRIAL: NCT06838663
Title: Comparative Outcomes of Robotic-Assisted Total Knee Arthroplasty: Cruciate-Retaining (CR) Versus Bi-Cruciate Stabilized (BCS) in a Randomized Controlled Trial
Brief Title: Robotic-Assisted Total Knee Arthroplasty: Cruciate-Retaining Versus Bi-Cruciate Stabilized
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024.599
Record Dates: First submitted 2025-02-19; First posted 2025-02-21 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty
Keywords: Knee Osteoarthritis; Knee OA; Total Knee Arthroplasty; Robotic-assisted TKA procedure
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Mastectomy, Segmental

STUDY DESIGN:
Masking Description: Subjects will be randomly assigned to robotic assisted Cruciate-Retaining (CR) or Bi-Cruciate Stabilized (BCS) TKA procedures groups according to a balanced randomization procedure using a 1:1 allocation ratio. To ensure balanced group assignment, a block randomization schedule will be generated. All subjects who sign the ICF and meet all inclusion and exclusion criteria will be randomized in a 1:1 randomization allocation ratio. The block size should be sufficiently small to allow approximately equal allocation of subjects in each group should the study be terminated prematurely whilst also being large enough so as the next treatment cannot be guessed. The study is non-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic assisted Cruciate-Retaining (CR) TKA procedures (Experimental): Patients who underwent Cruciate Retaining (CR) total knee arthroplasty (TKA)
  Interventions: Procedure: Robotic assisted Cruciate-Retaining (CR) TKA procedures
- Robotic assisted Bi-Cruciate Stabilized (BCS) TKA procedures (Experimental): Patients who underwent Bi-Cruciate Stabilized (BCS) total knee arthroplasty (TKA)
  Interventions: Procedure: Robotic assisted Bi-Cruciate Stabilized (BCS) TKA procedures

INTERVENTIONS:
Procedure: Robotic assisted Cruciate-Retaining (CR) TKA procedures — Patients who underwent Cruciate Retaining (CR) total knee arthroplasty (TKA)
  Arms: Robotic assisted Cruciate-Retaining (CR) TKA procedures
Procedure: Robotic assisted Bi-Cruciate Stabilized (BCS) TKA procedures — Patients who underwent Bi-Cruciate Stabilized (BCS) total knee arthroplasty (TKA)
  Arms: Robotic assisted Bi-Cruciate Stabilized (BCS) TKA procedures

SUMMARY:
The global prevalence of osteoarthritis of the knee with total knee arthroplasty performed is projected to substantially rise in the near future. This phenomenon is also observed in Hong Kong in which more than 4000 elective total joint replacement surgeries were performed in 2021 and over 30,000 patients are on the waiting list where some regions would have to wait for a median of more than 4 years. REAL INTELLIGENCE™ CORI™ (CORI Navigation) is a computer-assisted orthopedic surgical navigation and blurring system. CORI Navigation is designed to aid surgeons in planning and executing a procedure involving bone preparation for total knee arthroplasty (TKA) procedures. CORI Navigation is comprised of a console control unit, optical tracking camera, primary and secondary input displays (tablet and optional display monitor), and foot pedal. The CORI Navigation software consists of a patient and user management module, a surgical planner, and an intra-operative cutting module. Bi-Cruciate Stabilized (BCS) total knee arthroplasty (TKA) was designed for more kinematically functional implants that better reconstruct natural knee kinematics for activities of daily living. Surgical implant designs that resect the cruciate ligaments has emerged to simplify implantation and reduce surgical difficulty. The improvement of the biomechanical properties mimicking the natural kinematics of both the BCS and CR TKA may provide an effective solution to patient's dissatisfaction and impaired functional outcomes after surgery.

DETAILED DESCRIPTION:
Arthritis is a clinical syndrome of joint pain accompanied by varying degrees of functional limitation and reduced quality of life. Two common etiologies of arthritis are degeneration of the joint, osteoarthritis (OA), and inappropriate inflammatory response, rheumatoid arthritis (RA). OA is characterized by loss of cartilage, remodeling of adjacent bone, and inflammation in the affected joint. RA is a progressive inflammatory disease that eventually causes systemic joint damage and disability. Post-traumatic arthritis is a form of osteoarthritis following an injury to a joint. Inappropriate joint biomechanics due to deformities is the main risk factor for OA. The joint biomechanics are directly affected by the malalignment of the lower extremities due to anatomical deformities. Varus deformity is an excessive inward angulation of the lower leg and results in a bowlegged appearance. It may cause an overloading and cartilage wear in the medial knee compartment, which could support a degeneration of the knee joint leading to OA.

As of 2010, there were approximately 250 million people globally with osteoarthritis of the knee joint (3.6% of the global population). The prevalence was higher in females than in males. Initial treatment of arthritis may include physical therapy, nonsteroidal anti-inflammatory drugs (NSAIDs) such as ibuprofen and corticosteroids which can be taken orally or by injection.

Avascular necrosis (AVN) has several etiologies but fundamentally results from a decrease in blood flow to the affected bone, leading to cellular death. Studies have reported a 3.4% and 9.4% incidence of spontaneous osteonecrosis in persons older than 50 and 65 years of age, respectively. Initial treatment of AVN may include medication, stretching, and avoiding walking on the affected leg.

Complex epiphyseal fractures around the knee joint involve the distal femur or proximal end of the tibia. The management of these fractures, especially in elderly patients, is challenging. When the damage to the joint is advanced or available conservative treatment options are exhausted, knee arthroplasty is considered the most effective treatment for patients with any of these indications.

Total knee arthroplasty (TKA) is a highly successful and frequently performed surgical treatment to reduce disability caused by end-stage osteoarthritis and other conditions affecting articular cartilage. Technical outcomes for TKA are excellent, with favorable postoperative health-related quality of life. Also, survivorship of primary knee replacements is excellent with reported survivorship of 82.3% at 25 years. TKA has traditionally been indicated in the elderly population with relatively sedentary lifestyles, but more active, younger patients (<55) are receiving TKA due to the desire for a pain-free, active lifestyle with the demand projected to continue to increase for this group. A recent systematic review has shown that functional outcomes are similar in this population compared to elderly patients with no increase in the burden of revision.

In Australia, 660,000 primary TKAs have been performed in 2018. Since 2003, the number of knee replacement procedures undertaken has increased by 128%. The escalating prevalence of end-stage OA places an increased burden on healthcare providers, especially on less experienced surgeons and facilities that perform low numbers of arthroplasties. Lower volume hospitals (<25 procedures/year) report higher revision rates and more complications by 5 to 8 years compared to high volume hospitals (>200 procedures/year). Therefore, technology or techniques that could improve outcomes and reduce the risk of revision are becoming increasingly important.

Surgical factors that must be considered in knee arthroplasty include lower leg alignment, soft tissue balancing, maintenance of the joint line, and component size and fixation. Malalignment of components in any anatomical plane can cause major complications including aseptic loosening, instability, poor function, polyethylene wear, and pain. Additionally, implant malposition and malalignment of the joint can result in failure of the prosthesis. When not aligned within a narrow tolerance of ≤3° of the mechanical axis, poor functional outcomes, decreased implant survivorship, increased wear, and early failure from component loosening may occur.

Evidence has shown that neutral mechanical alignment provides optimal outcomes in knee arthroplasty, which is achieved with conventional alignment guides in approximately 75% of TKA cases. For partial knee procedures, approximately 30-60% of UKAs have been reported to be mal-aligned using conventional manual instruments. The importance of alignment can be demonstrated by observing higher revision rates of UKA attributed to malposition or malalignment of partial knees while roughly 25% of TKAs have been revised for instability or malalignment.

As an alternative to mechanical alignment, kinematic alignment technique for knee arthroplasty aims to restore the individual knee anatomy and ligament tension, to restore native knee kinematics. Kinematic alignment restores the obliquity and level of the joint line anatomically so the femoral component is slightly more valgus (1° to 2°) and the tibial component is slightly more varus (1° to 2°) than mechanically aligned components.

A significant innovation in knee arthroplasty has been the introduction of computer navigation and robotic-assisted surgery. One such technology is CORI. This system is a semi-autonomous image-free system. During the surgery, the surgeon maps the condylar landmarks and determines alignment indices to define the volume and orientation of bone to be removed. The tools to remove the bone and place the implants are controlled and manipulated by the surgeon with the guidance of a 3-dimensional digital map of the surgical surface.

Comparisons of navigation systems to conventional instruments have demonstrated that robotic platforms produce fewer positioning errors in both UKA and TKA. When used in medial or lateral UKA procedures, robotics reported short learning curves, increased accuracy in posterior tibial slope, and coronal tibial alignment in comparison to other alignment methods.

There are various total knee designs available in the market that promote their own benefits in restoring the natural kinematics of the knee to mimic the movement of the normal knee. Currently in our region, there are four commonly used robotic-assisted total knee arthroplasty designs available, which depend on the patient's factors and surgeon's preference. There is the Bi-Cruciate Retaining Total Knee Arthroplasty (BCR TKA), the Bi-Cruciate Stabilized Total Knee Arthroplasty (BCS TKA), the Posterior Stabilized Total Knee Arthroplasty (PS TKA), and the Cruciate Retaining Total Knee Arthroplasty (CR TKA).

The PS and BCS total knee arthroplasties are common choices as they sacrifice both the anterior cruciate ligament (ACL) and the posterior cruciate ligament (PCL) for simplification of implantation and reduction of surgical difficulty. The conventional PS TKA is a common feasible choice as it has shown long-term survivorship and acceptable patient outcomes. The BCS TKA similarly substitutes both the ACL and PCL but uses a unique dual cam-post mechanism to preserve normal knee kinematics and increase anterior-posterior stability throughout knee flexion.

On the other hand, preservation of the PCL in Cruciate Retaining (CR) total knee arthroscopy was traditionally believed to improve flexion and range of motion by restoring normal knee biomechanics and anatomical femoral rollback. PCL retention is also associated with better stairs performance, although the function of the PCL without the ACL is in debate. However, more recent studies have shown that there was a paradoxical anterior translation of the femur on the tibia during knee flexion, leading to the newer development of designs to retain both cruciate ligaments.

The Bi-Cruciate Retaining (BCR) total knee arthroplasty was designed for more kinematically functional implants that better reconstruct natural knee kinematics for activities of daily living by preserving both the anterior cruciate ligament (ACL) and the posterior cruciate ligament (PCL). BCR TKA historically has not been favored in the past due to its difficult surgical technique and complication rate, however, due to the recent emergence of new implant designs, it has gained back its popularity with improving functional outcomes and reducing complication rate. The ACL has been shown to be a factor for optimal knee kinematics and natural movement through its proprioceptive qualities. ACL deficient knees demonstrate posterior femoral position in full extension and increased medial femoral condyle translation during knee flexion. Preservation of both the ACL and PCL results in better flexion range, stability, and capacity to climb stairs.

On the other end of the spectrum, implant designs that resect the cruciate ligaments have emerged to simplify implantation and reduce surgical difficulty, such as the posterior cruciate retaining (PCR), posterior stabilized (PS), and the newer Bi-Cruciate Stabilized (BCS) total knee arthroplasty (TKA). In the normal knee, the lateral femoral condyle moves posterior across the tibial plateau with knee flexion, while the medial femoral condyle moves posterior in early flexion then anteriorly briefly before resuming posterior in the end of flexion. The BCS TKA is a convenient design that substitutes the sacrificed ACL and PCL with a unique dual cam-post mechanism to preserve normal knee kinematics and increase anterior-posterior stability throughout knee flexion.

The improvement of the biomechanical properties mimicking the natural kinematics of both the BCS and CR TKA may provide an effective solution to patient dissatisfaction and impaired functional outcomes after surgery. Therefore, an analysis of the knee kinematics of these patients with gait analysis, proprioception, and comparison of functional outcomes would aid the choice of implant.

Objective:

PRIMARY OBJECTIVE The primary objective of this study is to evaluate the use of CR and BCS in TKA procedure in achieving post-operative leg.

SECONDARY OBJECTIVE(S) The secondary objective of this study is to generate safety and performance evidence supporting the use of robotic assisted CR and BCS TKA procedures. To assess the safety and performance of robotic assisted CR and BCS TKA procedures up to 24 months after TKA surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a suitable candidate for a robotic-assisted TKA procedure
2. Subject requires a cemented TKA as a primary indication that meets any of the following condition:

   * Degenerative joint disease, including osteoarthritis
   * Rheumatoid arthritis
   * Avascular necrosis
   * Requires correction of functional deformity
   * Requires treatment of fractures that were unmanageable using other techniques
3. Subject is of legal age to consent and considered skeletally mature (≥ 18 years of age at the time of surgery)
4. Subject agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form), by signing the Ethical Committee (EC) or Institutional Review Board (IRB) approved informed consent form.
5. Subject plans to be available through two (2) year postoperative follow-up.
6. Applicable routine radiographic assessment is possible.

Exclusion Criteria:

1. Subject requires a TKA on the index joint as a revision for a previously failed surgery, or has the need for complex implants, or any other implant than a standard TKA (e.g. stems, augments, or custom made devices).
2. Subject has been diagnosed with post-traumatic arthritis.
3. Subject requires bilateral TKA.
4. Subject does not understand the language used in the Informed Consent Form.
5. Subject does not meet the indication or is contraindicated for TKA according to the specific Smith Nephew Knee System's Instructions For Use (IFU).
6. Subject has active infection or sepsis (treated or untreated).
7. Subject is morbidly obese with a body mass index (BMI) greater than 40.
8. Subject is pregnant or breast feeding at the time of surgery.
9. Subject, in the opinion of the Investigator, has advanced osteoarthritis or joint disease at the time of surgery and was better suited for an alternate procedure.
10. Subject has a condition(s) that may interfere with the TKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease, or an active, local infection).
11. Subject in the opinion of the Investigator has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, intellectual disability, drug or alcohol abuse.
12. Subject, in the opinion of the Investigator, has a neuromuscular disorder that prohibited control of the index joint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative leg alignment - Standard Radiographic Evaluation | pre-operatively and 6 weeks, 12 weeks，12months and 24 months after surgery
  The leg alignment should be measured from an antero-posterior (A/P) view standing weight bearing full leg ('long leg') x-ray. The following axes shall be identified:
  * Mechanical Axis of the femur: Axis from the center of the femoral head to the center of the distal femur.
  * Mechanical Axis of the tibia: Axis from the center of the proximal to the center of the distal tibia.
  Standard radiographic evaluation on antero-posterior (A/P) and lateral (L) views shall be performed 12&24 months after surgery in order to identify any radiographic observations such as radiolucent lines around the implant components. The presence of radiolucent lines, osteolysis & implant migration shall be recorded.

SECONDARY OUTCOMES:
2011 Knee Society Score | pre-operative visit and 6 weeks, 6 months, 12 months, and 24 months after surgery
  The 2011 KSS is a validated tool that combines an objective physician-derived component with a subjective subject-derived component. The 2011 KSS consists of 34 questions and provides sub-scores across 4 dimensions, including Objective Knee Score, Symptoms, Subject Satisfaction Score, Subject Expectation, and Functional Knee Score. The Objective Knee Score is rated by the clinician and assesses a range of clinical outcomes: TKA alignment, stability, range of motion (ROM) and symptoms. The Subject Satisfaction Score assesses the satisfaction with 5 daily activities (sitting, lying in bed, getting out of bed, light household duties, and leisure activities). The Subject Expectation Score evaluates the subject's expectations prior to surgery. The post-operative questions differ from the pre-operative questions and ask if the subject's pre-operative expectations have been met. As the pre- and post-operative scores are based on different questions, they cannot be directly compared.
Oxford Knee Score | pre-operative visit and 6 weeks, 6 months, 12 months and 24 months after surgery
  The Oxford Knee Score (OKS) is a Patient Reported Outcome (PRO) questionnaire that was developed to specifically assess the patient's perspective of outcome following Total Knee Arthroplasty. The OKS is a patient self-completion PRO containing 12 equally weighted questions on activities of daily living. The OKS has been developed and validated specifically to assess perceived function and pain answered on a Likert scale after TKA. Responses to each question ranges from 0-4 with a range of a possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome.
Forgotten Joint Score | pre-operative visit and 6 weeks, 6 months, 12 months, and 24 months after surgery
  The FJS comprises measures for the assessment of joint-specific patient reported outcomes. This questionnaire focuses on the study subject's awareness of the partially or fully replaced knee joint in everyday life. Joint awareness can be simply defined as any unintended perception of a joint. Subjects are asked to rate their awareness of their knee arthroplasty in 12 questions with a five point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale with a high value reflecting the ability of the subject to forget about the replaced knee joint during the activities of daily living.
Knee Injury and Osteoarthritis Outcome Score | pre-operative visit and 6 weeks, 6 months, 12 months, and 24 months after surgery
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury. The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life.
  The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved
The Western Ontario and McMaster Universities Osteoarthritis Index | pre-operative visit and 6 weeks, 6 months, 12 months, and 24 months after surgery
  The WOMAC is a widely used self-administered health status measure used in assessing pain, stiffness, and function in patients with OA of the hip or knee. It consists of three subscales: Pain: Measures the level of pain in the joint. Stiffness: Assesses the stiffness of the joint. Function: Evaluates the ability to perform daily activities such as walking, climbing stairs, and getting in and out of a chair. Minimum score: 0 (indicating no symptoms or functional limitations). Maximum score: 68 (for the original WOMAC scale, with higher scores reflecting greater severity of symptoms and limitations). Higher scores indicate worse outcomes, meaning more pain, more stiffness, and greater difficulty with daily activities. Lower scores suggest better joint health and function.
EQ-5D-5L | pre-operative visit as well as 6 weeks, 6- , 12 - and 24-months after surgery.
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system is used to describe the subject's health state and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems, and extreme problems. The subject is asked to indicate his/her health state by marking the most appropriate statement in each of the five areas.
  The EQ VAS records the subject's self-rated health on a vertical visual analogue scale. The endpoints on the scale are labelled "The best health you can imagine" and "The worst health you can imagine". The VAS can be used as a quantitative measure of health outcome as judged by the individual respondents.
Gait analysis | pre-operative visit as well as 6 weeks, 6- , 12 - and 24-months after surgery
  The biomechanical analysis will include gait cycle analysis, sit-to-stand, and stairs assessment. The analysis will be conducted with sixteen reflective markers being attached to specific anthropometric landmarks determined by the analysis software NEXUS 1.8.3 (VICON, Oxford Metrics Ltd., UK) and captured by sixteen infrared cameras. Initially the kinematic anatomical angles from the markers will be captured in a static trial using Vicon's Plug-In Gait model and then the patients will be asked to walk on an embedded force plate to measure the kinetic variables, including vertical and horizontal ground rection force and joint movements. The kinematic and kinetic variables will be processed and calculated in the Matlab (The Mathworks Inc., Natick, Massachusetts, USA). The patients will be asked to walk straight, climb up and down stairs a self-selected speed, and rise from sitting on a chair without using their arms.
Proprioception | pre-operative visit and 6 weeks, 6 months, 12 months, and 24 months after surgery
  The knee proprioception evaluation involved sensing of the joint position. An isokinetic dynamometer will be used in all of these procedures. All tests will be conducted with the patient in a seated position with the hip at approximately 90° and the entire back touching the backrest. The patient will be fixed to the seat by means of a belt.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication